CLINICAL TRIAL: NCT07291856
Title: Exploring the Impact of Dynamic Defocus Display Schemes on Ocular Health Indicators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: TREC2025-KY160
Record Dates: First submitted 2025-09-20; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-05

CONDITIONS: Visual Fatigue; Myopia
Keywords: Dynamic Defocus Display Technology; Visual Fatigue; visual function; Repeated Measures Design; Longitudinal Chromatic Aberration
MeSH Terms: conditions — Asthenopia; Myopia

STUDY DESIGN:
Intervention Model Description: This study is designed with a total of five groups, where participants will sequentially and randomly undergo all the intervention procedures.
Who Masked: Participant, Investigator
Masking Description: In this clinical trial, the masking is applied to the participants and the study staff who conduct the assessments. The participants are single-blinded, meaning they are unaware of the specific dynamic defocus mode they are assigned to during the trial. This is to ensure that their subjective responses, such as those recorded in the visual fatigue questionnaire, are not influenced by their knowledge of the intervention.
  The study staff who perform the assessments, including the measurement of critical flicker fusion frequency (CFF), accommodative function, and other ocular health indicators, are also blinded to the group assignments. This helps to prevent any potential bias in the data collection process, ensuring that the measurements are objective and reliable.
  The randomization sequence and group assignments are managed by a third-party institution, which maintains the integrity of the blinding. Only after all data have been collected and the initial analysis is complete will the bl
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control group (No Intervention): This group serves as the baseline comparison. Participants will perform the video-watching task on a conventional display with no intervention, allowing for the assessment of typical visual fatigue and ocular health indicators under standard conditions.
- Intervention Group A (Low defocus amplitude and high frequency) (Experimental): Participants will use a display with Dynamic Defocus Mode with low defocus amplitude and high frequency to perform a video browsing task. This group is designed with a specific dynamic defocus adjustment scheme, aimed at investigating the extent to which different dynamic defocus schemes can improve visual fatigue. Participants will be single-blinded to their group assignment. The intervention involves Dynamic Defocus Mode 1 and follows the VDT task protocol as designed in the trial.
  Interventions: Behavioral: Dynamic Defocus Mode
- Intervention Group B (low defocus amplitude and low frequency) (Experimental): Participants will use a display with Dynamic Defocus Mode with low defocus amplitude and low frequency to perform a video browsing task. This group is designed with a specific dynamic defocus adjustment scheme, aimed at investigating the extent to which different dynamic defocus schemes can improve visual fatigue. Participants will be single-blinded to their group assignment. The intervention involves Dynamic Defocus Mode 1 and follows the VDT task protocol as designed in the trial.
  Interventions: Behavioral: Dynamic Defocus Mode
- Intervention Group C (high defocus amplitude and high frequency) (Experimental): Participants will use a display with Dynamic Defocus Mode with high defocus amplitude and high frequency to perform a video browsing task. This group is designed with a specific dynamic defocus adjustment scheme, aimed at investigating the extent to which different dynamic defocus schemes can improve visual fatigue. Participants will be single-blinded to their group assignment. The intervention involves Dynamic Defocus Mode 1 and follows the VDT task protocol as designed in the trial.
  Interventions: Behavioral: Dynamic Defocus Mode
- Intervention Group D (high defocus amplitude and low frequency) (Experimental): Participants will use a display with Dynamic Defocus Mode with high defocus amplitude and low frequency to perform a video browsing task. This group is designed with a specific dynamic defocus adjustment scheme, aimed at investigating the extent to which different dynamic defocus schemes can improve visual fatigue. Participants will be single-blinded to their group assignment. The intervention involves Dynamic Defocus Mode 1 and follows the VDT task protocol as designed in the trial.
  Interventions: Behavioral: Dynamic Defocus Mode

INTERVENTIONS:
Behavioral: Dynamic Defocus Mode — Participants are required to complete a 50-minute video-watching task using a terminal display device that contains video content processed with different dynamic defocus modes. Specifically, participants will watch the same series of videos in different dynamic defocus modes. Participants will complete a total of 5 sets of video tasks (including the control group) in a random order.
  Arms: Intervention Group A (Low defocus amplitude and high frequency); Intervention Group B (low defocus amplitude and low frequency); Intervention Group C (high defocus amplitude and high frequency); Intervention Group D (high defocus amplitude and low frequency)

SUMMARY:
The present study is designed to explore the effects of dynamic defocus display technology on ocular health parameters using rigorous scientific approaches. It further examines the mechanisms through which this technology alleviates visual fatigue, thereby providing robust clinical evidence to support its practical application and widespread adoption.

DETAILED DESCRIPTION:
Research Content Recruit adults who meet the inclusion criteria and have long-term use of VDT (Visual Display Terminal) devices for the trial.

Compare the impact of different dynamic defocus modes on the visual fatigue symptoms of the subjects.

Analyze the mechanisms through which dynamic defocus modes alleviate visual fatigue.

Research Outcome Measures Primary Outcome Measures and Definitions Binocular Visual Function: A series of assessments of visual ability, including accommodative function (amplitude of accommodation, accommodative facility) and vergence function (near point of convergence, AC/A ratio).

Secondary Outcome Measures and Definitions Critical Flicker Fusion Frequency (CFF): To evaluate the degree of eye fatigue, with lower measured values indicating a higher degree of fatigue.

Visual Fatigue Questionnaire Score: To assess the subjective level of visual fatigue experienced by the subjects.

Refraction Results: To monitor changes in refractive status during the trial and evaluate the impact of different dynamic defocus modes on refractive state when using VDT devices at near distance.

ELIGIBILITY:
Inclusion Criteria:

Adults aged between 20 and 40 years, regardless of gender;

Refractive anisometropia ≤2.5D and corrected visual acuity of 1.0 or above in both eyes;

Habitual long-term use of electronic devices with LED light sources, such as computers and smartphones;

Currently not using any other blue light protection products or having ceased the use of such products for at least 2 weeks;

No known visually significant ophthalmic diseases;

Willing to participate in the trial and having signed the informed consent form.

Exclusion Criteria:

Abnormal accommodative function or other visual function abnormalities (e.g., strabismus, amblyopia);

Severe dry eye or history of ocular medication use;

Acute or chronic ocular surface inflammation, keratoconus, history of ocular surgery (e.g., refractive surgery), systemic diseases, or other conditions (e.g., wearing orthokeratology lenses and using atropine);

Photosensitivity, history of epilepsy, etc.;

Individuals unable to cooperate with the examination.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2025-08-20 (Actual); Primary Completion 2025-11-20 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Binocular Visual Function(amplitude of accommodation) | Baseline (before intervention), immediately after the 50-minute video-watching task for each of the five sessions, totaling ten completions per participant.
  The amplitude of accommodation refers to the maximum amount of accommodative power that the eye can exert to focus on near objects, typically measured in diopters.
Binocular Visual Function（accommodative facility） | Baseline (before intervention), immediately after the 50-minute video-watching task for each of the five sessions, totaling ten completions per participant.
  Accommodative facility, measured using a 2D flipper in cycles per minute (cpm), reflects the eye's ability to rapidly and efficiently change focus between near and far objects, indicating the dynamic functioning of the accommodative system.

SECONDARY OUTCOMES:
Critical Flicker Fusion Frequency(CFF) | Baseline (before intervention), immediately after the 50-minute video-watching task for each of the five sessions, totaling ten completions per participant.
  To evaluate the degree of eye fatigue, with lower measured values indicating a higher degree of fatigue.
Visual Fatigue Questionnaire Score | Baseline (before intervention), immediately after the 50-minute video-watching task for each of the five sessions, totaling ten completions per participant.
  The Computer Vision Syndrome Questionnaire (CVS-Q), which has been independently modified, comprises 16 response items. Participants will complete the questionnaire before and after the task to assess changes in ocular strain symptoms. By comparing the questionnaire scores obtained when using different dynamic defocus modes of the VDT devices, the effectiveness of dynamic defocus modes in alleviating subjective symptoms of ocular strain will be evaluated.
Refractive error status | Baseline (before intervention), immediately after the 50-minute video-watching task for each of the five sessions, totaling ten completions per participant.
  The refractive error status of the subjects was determined using a combination of automatic refractometer and subjective refraction, with results expressed in diopters.

OTHER OUTCOMES:
Optical Coherence Tomography Angiography | Baseline (before intervention), immediately after the 50-minute video-watching task for each of the five sessions, totaling ten completions per participant.
  Optical Coherence Tomography Angiography (OCTA) is a non-invasive imaging technique that provides detailed cross-sectional images of retinal and choroidal structures. It is particularly useful for evaluating the choroidal thickness, which can be measured precisely in micrometers.
Multispectral refraction topography | Baseline (before intervention), immediately after the 50-minute video-watching task for each of the five sessions, totaling ten completions per participant.
  Multispectral Refraction Topography (MRT) is an advanced imaging technique used to map the refractive properties of the eye across multiple wavelengths. By analyzing the eye's refractive profile at different spectral ranges, MRT offers a comprehensive understanding of the eye's optical characteristics.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospitol,Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No